CLINICAL TRIAL: NCT06363942
Title: A Personalized Video-based Exercise Program for Fall Prevention in Frail and Pre-frail Older Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jose Morais, Medical director, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-5973
Record Dates: First submitted 2024-03-15; First posted 2024-04-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Fall Injury; Frailty; Old Age; Atrophy; Age-Related Atrophy; Age-Related Sarcopenia
Keywords: frailty; exercise; older adult; ageing
MeSH Terms: conditions — Frailty; Atrophy; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE program (Experimental): Participants will be asked to carry out the SAFE program with the help of a caregiver. Our healthcare professionals will visit them during the first week to explain to them and their caregivers how to perform the exercises correctly while using our website. All exercises will be performed using video capsules available on our website (https://safe-seniors.com/fr). The exercises are divided into 4 levels of difficulty: level 1 (light); level 2 (moderate); level 3 (moderate to vigorous); and level 4 (vigorous). Each level lasts 25 to 30 minutes and includes 5 exercise categories split into 5 videos: warm-up, strength, balance, flexibility, and endurance. The exercise intervention will include 3 sessions per week over 12 weeks.
  Interventions: Other: SAFE program (exercise intervention)
- Control group (No Intervention): Participants will be asked to continue their activities of daily living without making any changes.

INTERVENTIONS:
Other: SAFE program (exercise intervention) — Participants will be asked to carry out the SAFE program with the help of a caregiver. Our healthcare professionals will visit them during the first week to explain to them and their caregivers how to perform the exercises correctly while using our website. All exercises will be performed using video capsules available on our website (https://safe-seniors.com/fr). The exercises are divided into 4 levels of difficulty: level 1 (light); level 2 (moderate); level 3 (moderate to vigorous); and level 4 (vigorous). Each level lasts 25 to 30 minutes and includes 5 exercise categories split into 5 videos: warm-up, strength, balance, flexibility, and endurance. The exercise intervention will include 3 sessions per week over 12 weeks.
  Arms: SAFE program

SUMMARY:
This is a randomized interventional clinical trial, whereby 100 participants will be randomized to either follow the SAFE exercise program (experimental group) or not (control group). At the end of the intervention, the experimental group will be encouraged to continue doing the exercises, and the control group will have the opportunity to participate in the SAFE exercises. 12 weeks post-intervention, the investigators will follow up with participants by telephone to follow up whether they are still following the SAFE program or not.

DETAILED DESCRIPTION:
For this study, the investigators will recruit 100 frail men and women aged 75 and over from the greater Montreal area. Enrolled participants will have 4 visits at their residence. The first visit, is a screening visit, the second is a pre-intervention assessment of cognition and functional abilities and explanation of the exercise program. The third visit will be a virtual visit, by phone call, and the final visit will be a post-intervention assessment of cognition and functional abilities.

Participants in the experimental group will engage in the SAFE exercises three times a week for 12 weeks at home while continuing their activities of daily living (ADLs) without any changes. Participants in the control group will not engage in the SAFE exercises but will be asked to maintain their ADLs without any changes. Before and after the 12-week intervention, all participants will complete a comprehensive battery of assessments to evaluate changes in their muscular strength, functional capacities, cognitive abilities and quality of life. At the end of the intervention, the experimental group will be encouraged to continue doing the exercises, and the control group will have the opportunity to participate in the SAFE exercises. 12 weeks post-intervention, the investigators will follow up with participants by telephone to follow up whether they are still following the SAFE program or not.

ELIGIBILITY:
Inclusion Criteria:

* Considered Frail or Pre frail according to Fried's criteria

Exclusion Criteria:

* Smoked within 6 months prior to study enrollment,
* dementia diagnosos,
* Abused drugs, medication or alcohol within up to 30 days prior to the start of the study.
* drug or alcohol-addiction,
* Heart disease, history of heart attacks or electrocardiogram abnormalities
* Any family history of thrombosis, thrombosis risk,
* hypocalcaemia,
* uric acidemia,
* orthostatic intolerance,
* vestibular disorders,
* considerable musculoskeletal issues,
* chronic back pain,
* head trauma,
* seizures,
* ulcers,
* renal stones,
* gastro-esophageal reflux disease,
* renal function disorder,
* hiatus hernia,
* migraines,
* mental illness diagnosis
* prescribed medication that may interfere with the interpretation of the results

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective 1 | 12 weeks
  Number of participants that displayed changes on their functional testing (SPPB) in comparison with their baseline and the control group after having participated in the SAFE program, following the 12 week intervention.
Objective 2 | 12 weeks
  Number of participants that displayed changes on their cognitive (STROOP) in comparison with their baseline and the control group after having participated in the SAFE program, following the 12 week intervention.

SECONDARY OUTCOMES:
Objective 4 | 12 weeks
  Number of participants that displayed changes on their FES-I test in comparison with their baseline and the control group after having participated in the SAFE program, following the 12 week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Morais, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital - Glen site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of the study.

REFERENCES:
- [Background] Masud T, Morris RO. Epidemiology of falls. Age Ageing. 2001 Nov;30 Suppl 4:3-7. doi: 10.1093/ageing/30.suppl_4.3. No abstract available. PMID 11769786
- [Background] Al-Aama T. Falls in the elderly: spectrum and prevention. Can Fam Physician. 2011 Jul;57(7):771-6. PMID 21753098
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Sherrington C, Tiedemann A, Fairhall N, Close JC, Lord SR. Exercise to prevent falls in older adults: an updated meta-analysis and best practice recommendations. N S W Public Health Bull. 2011 Jun;22(3-4):78-83. doi: 10.1071/NB10056. PMID 21632004
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Jensen AR, Rohwer WD Jr. The Stroop color-word test: a review. Acta Psychol (Amst). 1966;25(1):36-93. doi: 10.1016/0001-6918(66)90004-7. No abstract available. PMID 5328883